CLINICAL TRIAL: NCT04221607
Title: An Intimacy Intervention for Couples Completing Breast or Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Keitner/Family Therapy Research Grant (Unknown)
Responsible Party: Principal Investigator, Don Dizon, Professor of Medicine, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1413727
Record Dates: First submitted 2020-01-04; First posted 2020-01-09 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Sexual Dysfunction; Breast Cancer; Prostate Cancer
Keywords: intimacy; sensate focus; survivorship; breast cancer; prostate cancer
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Feasibility of intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility (Experimental): Sensate Focus Exercises aim to help couples be more present with one another through talking and through touch.
  Interventions: Other: Sensate Focus exercise

INTERVENTIONS:
Other: Sensate Focus exercise — Structured exercise to enhance intimacy

SUMMARY:
This project seeks to help patients address and improve intimacy at the end of treatment for breast or prostate cancer. It is intended to address the needs of cancer survivors, broadly defined as paftients and their loved ones or caregivers facing a cancer diagnosis. While we know sexual health is impacted by the diagnosis and treatments for cancer, we also are increasingly aware that partners and spouses are also impacted by the experience. Yet, there are no evidence based interventions that focus on the couple's recovery after the initial cancer experience.

The objective of this study is to look at the impact of an intimacy intervention at the completion of cancer treatment for couples facing breast or prostate cancer. We will enroll patients and their intimate partners in this study in two phases. In the first phase, couples will receive sensate focus homework, explained to them at a standard survivorship care visit (SCV) by a study nurse practitioner (NP). The objective in the first phase is to see if this is something feasible by looking at how many use sensate focus homework in 6 weeks. If it is not feasible, we will rework the study based on what we learned. However, if it is feasible, we will reopen the study to a larger group and employ a random assignment to an SCV with or without sensate focus homework. This phase will give us evidence of efficacy that we will use to propose a larger randomized trial, potentially in the National Cancer Institute system.

Participants will be asked to answer questionnaires at baseline, 6 weeks, and then at 12 weeks during phase 2. Those who complete treatment at 12 weeks will be re-contacted 6 months after protocol enrollment for an optional end of treatment interview to assess what they thought of the intervention, including sensate focus homework itself and the timing.

DETAILED DESCRIPTION:
The National Comprehensive Cancer Network (NCCN) identifies sexual dysfunction as a major issue facing cancer survivors (defined broadly as patients and their caregivers, starting at the point of the index cancer diagnosis). It is well known that a cancer diagnosis and treatment negatively impacts partner relationships and quality of life (QOL) (for both patient and partner). Despite this, only about a third of patients seek assistance, and the figures regarding assistance from caregivers is lacking.

The etiology of sexual dysfunction is multifactorial and includes problems with sexual desire and pleasure, hormonal deficiencies, vaginal and penile alterations related to treatment, delayed or absent orgasm and/or ejaculation, pain with intercourse, erectile dysfunction, and psychological problems such as anxiety, depression, and changes in body-image. Unfortunately, interventions have largely focused on ways to improve sexual function, although even these are limited. Additionally, clinicians are often reluctant to address sexual function with their patients due to their lack of training and discomfort in engaging in these conversations. Given the well-documented burden of sexual dysfunction, there is a compelling need to develop interventions to address sexual health, for both patient and partner while encouraging clinicians to discuss sexual health issues.

Beyond the issues of the individual, couples and families are also impacted by cancer treatment. A wide body of literature shows that a cancer experience can add additional demands on couples, especially in the realms of communication, intimacy, and sexuality. A small study of 8 couples where the female partner had breast cancer identified three themes of significance: (1) disconnection from the relationship, due to the woman prioritizing her own needs before those of the partner or of them as a couple; (2) renegotiation of the couple relationship; and (3) need for support for negotiating going forward as a couple. Unfortunately, they also comment on the limited evidence-based interventions to aide this transition, particularly for the couple.

In this project, the investigators will build upon standard procedures to address intimacy at the end of curative intent therapy through sensate focusing exercises (SF). SF will be delivered during a face-to-face survivorship visit using a trial-specific script.

The project will proceed in two phases. During phase 1, the investigators will assess feasibility by conducting a prospective pilot study. During phase 2, the investigators will conduct a randomized trial comparing survivorship care with or without sensate focusing.

This project has the potential to substantially enhance the care of survivors. By implementing such an intervention to improve sexual function, we aim to enhance the QOL and intimacy of cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) with histologically proven breast or prostate cancer
* Ability to speak English or able to complete questionnaires with assistance required from an interpreter or family member.
* Completed curative intent treatment for cancer no more than 6 months prior to study enrollment. Treatment may have consisted of surgery, chemotherapy, and/or radiation therapy. Patients on extended adjuvant (maintenance) treatment will be allowed to enroll.
* In a stable non-married relationship or otherwise partnered or married.
* Partner willing to participate in study

Exclusion Criteria:

* history of significant psychiatric or other co-morbid disease, which the treating clinician believes prohibits the patient's ability to participate in the informed consent procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Phase one: Feasibility | Four weeks
  Proportion of couples enrolled in phase one who are practicing sensate focus at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Don S Dizon, MD, Principal Investigator — Rhode Island Hospital
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No